CLINICAL TRIAL: NCT07318857
Title: Clinical Investigation of the Transfer Accuracy of Semi-Digital and Fully Digital Indirect Bonding Trays
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Selcuk University (Other)
Responsible Party: Principal Investigator, Ramazan Emre Karakoç, Principal Investigator, Selcuk University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SU-ORTO-2542
Record Dates: First submitted 2025-12-15; First posted 2026-01-06 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-12

CONDITIONS: Indirect Bonding

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Semi-Digital Transfer Tray Group (Active Comparator): Indirect bonding using transfer trays prepared by thermoforming over 3D printed models
  Interventions: Procedure: Semi-Digital Indirect Bonding
- Fully Digital Transfer Tray Group (Experimental): Indirect bonding using directly 3D printed transfer trays designed in CAD software
  Interventions: Procedure: Fully Digital Indirect Bonding

INTERVENTIONS:
Procedure: Semi-Digital Indirect Bonding — Bonding brackets using thermoformed transfer trays.
  Arms: Semi-Digital Transfer Tray Group
Procedure: Fully Digital Indirect Bonding — Bonding brackets using 3D printed transfer trays.
  Arms: Fully Digital Transfer Tray Group

SUMMARY:
This randomized clinical study compares the transfer accuracy of semi-digital and fully digital indirect bonding trays in orthodontic treatment. Thirty-two patients were randomly divided into two groups to receive brackets bonded with either semi-digital trays (thermoformed on 3D printed models) or fully digital trays (directly 3D printed). The primary outcome measures are linear and angular deviations between the virtually planned and actual clinical bracket positions, analyzed using 3D superimposition techniques.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 12-25 years in permanent dentition
* Had a mild irregularity (≤ 3mm)
* Requiring comprehensive fixed orthodontic treatment and had no previous orthodontic therapy
* Not having malformed, excessively rotated, large restorations or missing teeth in the upper arch

Exclusion Criteria:

* Inadequate oral hygiene
* Had severe crowding
* Systemic or craniofacial anomalies

Ages: 12 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 32 (Actual)
Dates: Start 2023-06-15 (Actual); Primary Completion 2024-05-21 (Actual); Study Completion 2024-06-24 (Actual)

PRIMARY OUTCOMES:
Linear Transfer Accuracy | Immediately after the bonding procedure (Day 1)
  Linear deviations between the virtually planned bracket positions and the actual clinical bracket positions. Measurements are calculated by superimposing the post-bonding intraoral scans onto the virtual setup models using GOM Inspect software.
  Unit of Measure: Millimeters
Angular Transfer Accuracy | Immediately after the bonding procedure (Day 1)
  Angular deviations between the virtually planned bracket positions and the actual clinical bracket positions. Measurements are calculated by superimposing the post-bonding intraoral scans onto the virtual setup models using GOM Inspect software.
  Unit of Measure: Degrees

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Orthodontics, Faculty of Dentistry, Selcuk University, Konya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided